CLINICAL TRIAL: NCT02062034
Title: Efficacy of Ubiquinone and Combined Antioxidant Therapy on Progression, Oxidative Stress Markers and Mitochondrial Dysfunction in Non-proliferative Diabetic Retinopathy: A Phase 2a Randomized Double-blind Placebo-controlled Study
Brief Title: Efficacy of Ubiquinone and Combined Antioxidant Therapy in Non-proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Alejandra Guillermina Miranda Diaz, PhD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDNP-20100102
Record Dates: First submitted 2013-07-17; First posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Non-proliferative Diabetic Retinopathy; Diabetes Mellitus Type 2
Keywords: Oxidative stress; Mitochondrial dysfunction; Ubiquinone; Antioxidant combined therapy; Diabetic retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Mitochondrial Diseases; Diabetic Retinopathy | interventions — Ubiquinone; coenzyme Q10; Lutein; Zeaxanthins; astaxanthine; Ascorbic Acid; Vitamin E; Zinc; Copper

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ubiquinone (Experimental): 400mg daily of oral ubiquinone for 24 weeks
  Interventions: Drug: Ubiquinone
- Combined antioxidant therapy (Experimental): (1mg copper + 20mg zinc + 180mg vitamin C + 30mg vitamin E + 1mg zeaxanthin + 4mg astaxanthin + 10mg lutein) daily of oral antioxidant combined therapy for 24 weeks
  Interventions: Drug: Combined antioxidant therapy
- Placebo (Placebo Comparator): Placebo. 100mg daily oral intake for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ubiquinone — 400mg daily of oral ubiquinone for 24 weeks
  Other Names: coenzyme Q10
  Arms: Ubiquinone
Drug: Combined antioxidant therapy — (1 mg copper, 20 mg zinc, 180 mg vitamin C, 30 mg vitamin E, 1 mg zeaxanthin, 4 mg astaxanthin, 10 mg lutein) daily of oral, all of them in one Tablet for 24 weeks
  Other Names: lutein; zeaxanthin; astaxanthin; vitamin C; vitamin E; zinc; copper
  Arms: Combined antioxidant therapy
Drug: Placebo — 100 mg of oral placebo with identical appearance, form, size than ubiquinone and antioxidant combined therapy for 24 weeks
  Other Names: Inactive drug
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of ubiquinone and combined antioxidant therapy on progression, clinical regression, oxidative stress markers and mitochondrial dysfunction in non-proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
The investigators are interested in demonstrating the efficacy of Ubiquinone and combined antioxidant therapy in the pharmacological management of diabetic retinopathy since early stages.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus
* Patients with non proliferative diabetic retinopathy
* Glycated hemoglobin < 12.0%
* Signing of informed consent

Exclusion Criteria:

* Patients with clinically significant macular edema
* Patients with diabetic retinopathy advanced lesions that have required or require specific treatment (laser, vitrectomy)
* Pretreatment with argon laser or excimer laser Ophthalmology surgery
* Any other associated ocular pathology (glaucoma, cataracts, changing cornea dystrophy, macular degeneration)
* Pregnancy, lactation, inadequate use of contraception
* Antioxidant drug and/or supplements six months previous to enrollment
* Renal and/or hepatic failure
* Age under 30 or over 75 years
* Severe cardiovascular disease (myocardial infarction, stroke, severe peripheral vasculopathy)
* Blood dyscrasias
* Have or have had cancer or other serious illness
* Neurodegenerative process
* Allergy to vitamins

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Oxidative Stress markers | 24 weeks
  In this study the oxidative stress markers are composed of lipid peroxidation, nitric oxide, erythrocyte glutathion peroxidase activity, erythrocyte catalase activity, total antioxidant capacity and erythrocyte membrane fluidity.
  * Lipid peroxidation (baseline and final values) given as malondialdehyde (MDA) and 4-hydroxyalkenals (4HDA) expressed in μmol/L
  * Nitric oxide (NO) Levels of the NO catabolites nitrites/nitrates expressed in pmol/mL (baseline and final values)
  * Erythrocyte glutathion peroxidase activity measured in U/min/mg protein (baseline and final values)
  * Erythrocyte catalase activity expressed in U/mg protein (baseline and final values)
  * Total antioxidant capacity measured in milliequivalent/mL (baseline and final values)
  * Erythrocyte membrane fluidity, calculated using the fluorescence ratio of the excimer (Ie) to monomer (Im). The Ie/Im ratio.

SECONDARY OUTCOMES:
Mitochondrial dysfunction markers | 24 weeks
  In this study the mitochondrial dysfunction markers are composed of hydrolysis of adenosine triphosphate and membrane fluidity in submitochondrial particles of platelets.
  * Hydrolysis of adenosine triphosphate: The hydrolytic activity of mitochondrial F0/F1-ATPase (F0/F1-adenosine triphosphatase) was measured as the liberation of inorganic phosphate from platelet mitochondria. Expressed in nmol of phosphate. Baseline and final values.
  * Membrane fluidity in submitochondrial particles of platelets. Calculated usig the fluorescence ratio of the excimer (Ie) to monomer (Im). The Ie/Im ratio. (Baseline and final values)
Progression and regression of non-proliferative diabetic retinopathy | 24 weeks
  Evaluated with International clinical diabetic retinopathy disease severity scale, fluorescein angiography and color fundus photographs.
  Baseline and final stage.

OTHER OUTCOMES:
Security profile | 24 weeks
  In this study the security profile markers are composed of intraocular pressure, visual acuity, renal function, and liver profile.
  Intraocular pressure. expressed in mmHg (baseline and final values) Visual acuity measured in decimal scale (baseline and final values) Renal function: serum urea (mg/dL), serum creatinine (mg/dL). (Baseline and final values) Liver profile: total serum bilirubin (mg/dL), indirect bilirubin (mg/dL), direct bilirubin (mg/dL) (Baseline and final values).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra G. Miranda-Díaz, PhD, Study Director — University of Guadalajara; José A. Castellanos-González, M.Sc., Study Chair — University of Guadalajara; Adolfo D. Rodriguez-Carrizalez, M.Sc., Study Chair — University of Guadalajara
Locations (1):
- Cardiovascular Research Unit, University of Guadalajara, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Result] Hernandez-Ojeda J, Cardona-Munoz EG, Roman-Pintos LM, Troyo-Sanroman R, Ortiz-Lazareno PC, Cardenas-Meza MA, Pascoe-Gonzalez S, Miranda-Diaz AG. The effect of ubiquinone in diabetic polyneuropathy: a randomized double-blind placebo-controlled study. J Diabetes Complications. 2012 Jul-Aug;26(4):352-8. doi: 10.1016/j.jdiacomp.2012.04.004. Epub 2012 May 16. PMID 22595020
- See also: The effect of rosuvastatin in Diabetic Polyneuropathy: A Phase 2a Randomized Double-blind Placebo-controlled Study — http://clinicaltrials.gov/ct2/show/record/NCT01622777